CLINICAL TRIAL: NCT04003233
Title: Limited-efficacy Testing of Spring Distraction System (SDS) and Unilateral One-way Rod (MID-C) for Early Onset Scoliosis
Acronym: UniPOWR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the termination of the collaboration of ApiFix ltd. and the UMC Utrecht
Sponsor: UMC Utrecht (Other)
Collaborators: Apifix (Industry)
Responsible Party: Principal Investigator, M.C. Kruyt, MD, PhD, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL63511.041.17
Record Dates: First submitted 2019-06-07; First posted 2019-07-01 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Early-Onset Scoliosis Deformity of Spine (Disorder); Idiopathic Scoliosis
Keywords: Growth friendly system; Distraction system; Early Onset Scoliosis; Unilateral

STUDY DESIGN:
Intervention Model Description: Participants will be randomized and assigned to either SDS or MID-C.
Who Masked: Participant
Masking Description: Participants are blinded to the medical device till the surgery. After the surgery participants are able to see which medical device is implanted on X-rays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spring Distraction System (Experimental): The SDS device will be implanted during a scoliosis correction operation.
  Interventions: Device: SDS
- Minimal Invasive Deformity Correction system (Experimental): The MID-C device will be implanted during a scoliosis correction operation.
  Interventions: Device: MID-C

INTERVENTIONS:
Device: SDS — The SDS will be added to a traditional growing rod (TGR) of 4.5 or 5.5mm.
  Arms: Spring Distraction System
Device: MID-C — The MID-C system consists of a unilateral one-way ratchet rod that is connected to the spine with polyaxial connectors
  Arms: Minimal Invasive Deformity Correction system

SUMMARY:
The primary aim of this study is to investigate the limited efficacy of these innovative surgical solutions in treatment of Early Onset Scoliosis (EOS) in terms of maintaining reduction while maintaining spinal growth. The secondary aim is to compare both devices for these and other parameters as well as safety.

DETAILED DESCRIPTION:
Rationale: EOS is a severe and potentially life-threatening disorder since a disturbance of spinal development leads to impaired development of the trunk, with cardio-respiratory failure as a result, often early in adult life. Several innovative solutions have been developed to treat growing children with severe EOS. The SDS device was developed internally at the dpt. of orthopedics at the UMC Utrecht, the Netherlands, the MID-C device was developed by the company ApiFix Ltd.

Objective: The primary aim of this study is to investigate the limited efficacy of these innovative surgical solutions in treatment of early onset scoliosis in terms of maintaining reduction while maintaining spinal growth. The secondary aim is to compare both devices for these and other parameters as well as safety.

Study design: A feasibility study using two prospective cohorts according to an open label randomized clinical trial (RCT) design. The study will be done in two tertiary referral centers (UMC Utrecht and Amsterdam UMC). Primary endpoints are maintenance of curve correction as well as complications. These data will be compared to a recently described cohort of patients that received a "standard treatment" (Magnetically controlled growing rod (MCGR)). The same endpoints as well as secondary outcomes, will be compared between the two new treatments.

Study population: Children with idiopathic(-like) early onset scoliosis with an indication for a growing rod implant.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant skeletally immature children, 6-12 yrs. of age, with open triradiate cartilages on X-ray
* Scoliosis diagnosis prior to the age 10
* Diagnosis of idiopathic or mild syndromic scoliosis (e.g. 22q11DS, Trisomy 21 or 9, Coffin-Siris)
* Progressive scoliosis qualified for growth system surgery
* One curve for treatment with an apex below Th5 and a proximal end vertebra below Th2
* The primary curve must be between 35 and 75 degrees coronal Cobb angle
* The primary curve must be non-rigid (i.e. the curve reduces on bending X-rays to <35 degrees or reduces >30% )
* Normal or hypokyphotic sagittal alignment (Th5 -Th12 < 50 degrees) on lateral X-rays

Exclusion Criteria:

* Patients with an obvious neuromuscular disease
* Patients that are severely mentally retarded
* Patients with a scoliosis that extends to the pelvis or the cervicothoracic region
* Patients with a main curve of more than 8 vertebra Cobb to Cobb
* Patients with a skeletal dysplasia that effects growth (e.g. achondroplasia, SED)
* Patients with a systemic disease which severely influences bone quality (e.g. osteogenesis imperfecta, metabolic diseases)
* Patients with soft tissue weakness (e.g. Ehler Danlos, Marfan, Neurofibromatosis, Prader Willi)
* Patients with an active systemic disease such as Juvenile Idiopathic Arthritis, HIV or oncologic treatment
* Patients with a previous surgical fusion of the spine

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Limited-efficacy of SDS and MID-C in terms of curve correction maintenance: changes in cobb angle | Until 1 year post-operative FU
  changes in cobb angle on radiographs post-op and at 4 weeks, 3 months and 12 months follow-up (FU). A maximum of 5 degrees increase will be the threshold to define maintenance.
Incidence of Treatment-Emergent Serious Adverse Events of SDS and MID-C | Until 1 year post-operative FU
  Reported treatment related Serious Adverse Events (SAEs) per-operatively and at 4 weeks, 3 months and 12 months FU.

SECONDARY OUTCOMES:
Limited-efficacy of SDS and MID-C in terms of spinal length | Until 1 year post-operative FU
  Changes in length of T1-T12, T1-S1 and the instrumented segment in mm on calibrated Anterior Posterior (AP) X-rays post-op and at 4 weeks, 3 months and 12 months FU.
SDS vs. MID-C with respect to limited-efficacy in terms of curve correction maintenance | Until 1 year post-operative FU
  changes in cobb angle on radiographs post-op and at 4 weeks, 3 months and 12 months FU. A maximum of 5 degrees increase will be the threshold to define maintenance.
SDS vs. MID-C with respect to limited-efficacy in terms of spinal length | Until 1 year post-operative FU
  Changes in length of T1-T12, T1-S1 and the instrumented segment in mm on calibrated AP X-rays post-op and at 4 weeks, 3 months and 12 months FU.
SDS vs. MID-C with respect to the incidence of Treatment-Emergent Serious Adverse Events | Until 1 year post-operative FU
  Reported treatment related SAEs per-operatively and at 4 weeks, 3 months and 12 months FU.
SDS vs. MID-C with respect to surgery time | Until 1 year post-operative FU
  Surgery time in minutes
SDS vs. MID-C with respect to blood loss during surgery | Until 1 year post-operative FU
  blood loss in cc
SDS vs. MID-C with respect to length of hospital stay | Until 1 year post-operative FU
  length of hospital stay in days
SDS vs. MID-C with respect to recovery time | Until 1 year post-operative FU
  recovery time in minutes
SDS vs. MID-C with respect to bone density | Until 1 year post-operative FU
  Bone density changes of the bypassed vertebrae on Dual Energy X-ray Absorptiometry (DEXA)scan post-op and at 3 months en 12 months FU.
SDS vs. MID-C with respect to Quality Of Life (QOL) on the Early Onset Scoliosis Questionnaires (EOSQ-24) | Until 1 year post-operative FU
  Parent reported QOL and performance is assessed with the 24-item Early Onset Scoliosis Questionnaires (EOSQ-24) pre-op and at 4 weeks, 3 months and 12 months FU. EOSQ-24 covers the following domains: Child's Health Related Quality of Life (16 items), Family Impact (2 items) and Satisfaction (2 items).
SDS vs. MID-C with respect to flexibility of the spine | Until 1 year post-operative FU
  Flexibility and 3D rotation of the spine on dynamic echography (Scolioscan)
SDS vs. MID-C with respect to 3D development of the spine | Until 1 year post-operative FU
  Apical Vertebral Rotation based on MRI
SDS vs. MID-C with respect to patient appearance | Until 1 year post-operative FU
  sagittal balance on clinical photographs post-op and at 1 year FU

CONTACTS AND LOCATIONS:
Overall Officials: Moyo C Kruyt, MD, PhD, Principal Investigator — UMC Utrecht
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam, North Holland
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No